CLINICAL TRIAL: NCT05021419
Title: Efficacy of a Streamlined Heart Failure Optimisation PRoTocol for Patients with Severely Impaired Left Ventricular Systolic Function, a Randomised Controlled Trial (SHORT Trial)
Brief Title: Efficacy of a Streamlined Heart Failure Optimization Protocol
Acronym: SHORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Queen Elizabeth Hospital King's Lynn NHS Foundation Trust (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Qehkl
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure with Reduced Ejection Fraction; Chronic Heart Failure
Keywords: Medication Sequencing; Optimization
MeSH Terms: interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Arm (Active Comparator): Both the current European Society of Cardiology (ESC) and the National Institute of Health and Care Excellence (NICE) guidelines advise that chronic stable heart failure patients with severely impaired left ventricular systolic function should initially be optimized as follows:
  Visit 1: Angiotensin-converting enzyme inhibitor (ACEi)/Angiotensin receptor blocker (ARB) and Low dose Beta blocker commenced Visit 2: ACEi/ARB up-titrated; (Beta Blocker up-titrated) Visit 3: ACEi/ARB up-titrated; (Beta Blocker up-titrated) Visit 4: Mineralocorticoid receptor antagonist (MRA) added Visit 5: MRA up-titrated Visit 6: Switch ACEi/ARB to Entresto 49/51 mg twice daily (BD) Visit 7: Modify Entresto dose to 97/103 mg BD Visit 8: Sodium-glucose cotransporter-2 inhibitor (SGLT2i) started
  Interventions: Other: Standard Protocol
- Streamlined protocol arm (Experimental): Patients are optimized according to the accelerated protocol adapted from and based on the principles proposed by Prof McMurray and Prof Packer (Circulation 2021;143:875-877)
  Visit 1: Low dose Beta Blocker started, SGLT2i started & Entresto* started
  *The starting dose of Entresto will be determined by the baseline blood pressure (BP) (a dose of 24/26 mg twice daily (BD) is to be started if the systolic BP is less than 110 mmHg otherwise a dose of 49/51 mg BD is to be started)
  Visit 2: MRA added if renal function and potassium levels permit (Beta Blocker increased if BP and pulse rate permit)
  Visit 3: MRA/Entresto up-titrated if BP and renal function and potassium levels permit (Beta Blocker increased if BP and pulse rate permit)
  Visit 4+: Beta Blocker increased if BP and pulse rate permit. Further visits may be required to facilitate a gentle up-titration of Beta Blockers.
  Interventions: Other: Streamlined protocol

INTERVENTIONS:
Other: Streamlined protocol — A streamlined drug protocol for optimizing heart failure medication
  Arms: Streamlined protocol arm
Other: Standard Protocol — Current standard optimization protocol as per NICE and ESC
  Arms: Standard Arm

SUMMARY:
The SHORT trial compares the current standard optimization protocol to a shortened protocol in a randomized control trial.

DETAILED DESCRIPTION:
The SHORT trial compares the current standard optimization protocol to a shortened protocol in a randomized control trial. It assesses whether an accelerated protocol leads to faster optimization and a greater degree of optimization.

ELIGIBILITY:
Inclusion Criteria:

* Ejection fraction of less than or equal to 40%
* Increased NT-proBNP level:
* ≥ 600 pg per milliliter or
* ≥400 pg per milliliter if they had been hospitalized for heart failure within the previous 12 months or
* patients with atrial fibrillation or atrial flutter on baseline electrocardiography were required to have an NT-pro BNP level of at least 900 pg per milliliter, regardless of their history of hospitalization for heart failure or
* recent heart failure admission or clinical diagnosis of heart failure.
* Patients who are either naïve to or taking no more than 25% target doses of Beta Blockers or ACEi or ARB before starting the trial.

Exclusion Criteria:

* Systolic BP of less than 100 mmHg on 2 consecutive measurements
* Estimated glomerular filtration rate (eGFR) less than 30 ml/min/1.73m2
* Type 1 diabetes mellitus
* Cognitive impairment that in the opinion of the investigator may lead the patient to be unable to understand and/or comply with the study medications, procedures and/or follow-up
* Uncorrected primary valvular disease
* Active malignancy treatment at time of visit 1
* Women of child-bearing potential who are not willing to use a medically accepted method of contraception that is reliable in the judgement of the investigator*
* Women who are pregnant or breastfeeding
* History of angioedema, or hereditary or idiopathic angioedema
* Severe hepatic impairment, biliary cirrhosis or cholestasis
* Patients who are receiving treatment with an aliskiren-containing product who have diabetes mellitus or renal impairment (eGFR <60 ml/min/1.73 m2)

  * Highly effective methods of contraception include implants, injectables, combined oral contraceptives (the participant must have been on a stable dose for at least 3 months before entering the trial), intrauterine device, vasectomised partner, or true sexual abstinence (when this is the preferred and usual lifestyle of the patient and does not include periodic abstinence [e.g. calendar, ovulation, symptothermal or post-ovulation methods]). Use of such methods must be maintained throughout the trial and for 7 days after the end of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-17 (Actual); Primary Completion 2024-01-07 (Actual); Study Completion 2024-01-07 (Actual)

PRIMARY OUTCOMES:
Time to point of optimization | Maximum follow-up 6 months
  Do patients on the streamlined protocol reach the point of optimization* earlier?
  *point of optimization is defined as the point in time at which no medication could be increased further either due to achievement of target doses or limited by symptoms, low heart rate, BP, or raised serum potassium or serum Creatinine.

SECONDARY OUTCOMES:
Degree of optimization reached | Maximum follow-up 6 months
  1. Do patients on the streamlined protocol reach a greater "degree of optimization" **?
  **degree of optimization is defined as the average percentage of the target doses reached across the four heart failure drug groups at the point of optimization.
Number of appointments required | Maximum follow-up 6 months
  Do patients on the streamlined protocol require fewer appointments to reach the point of optimization?
Number of Complications | Maximum follow-up 6 months
  Is the streamlined protocol as safe as the current best practice protocol? The number of symptomatic hypotension requiring hospitalization and hyperkalaemia requiring hospitalization.
Change in NT-pro BNP | 6 months
  Do patients on the streamlined protocol have a greater decrease in N-terminal pro-B-type natriuretic peptide (NT-pro BNP) levels 6 months after the initial optimization appointment?
Symptomatic change | 6 months
  5. Do patients on the streamlined protocol have a greater reduction in symptoms at 6 months after the initial optimization appointment? Use of the Kansas City Cardiomyopathy Questionaire score***.
  ***Kansas City Cardiomyopathy Questionaire score assesses health status of patients with heart failure via four domains: Physical Limitation, Symptom Frequency, Quality of Life and Social Limitations. Each domain provides an individual score from 0 to 100, with 0 denoting the worst and 100 the best possible health status.
Composite of cardiovascular death and worsening heart failure | 6 months
  Do patients on the streamlined protocol have a lower incidence of the composite endpoint of cardiovascular death and worsening heart failure (defined as hospitalization or an urgent visit resulting in intravenous therapy for heart failure)?

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf M Duehmke, BSc MBBS PhD, Principal Investigator — The Queen Elizabeth Hospital King's Lynn NHS Foundation Trust
Locations (1):
- Queen Elizabeth Hospital King's Lynn, Kings Lynn, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Guideline Centre (UK). Chronic Heart Failure in Adults: Diagnosis and Management. London: National Institute for Health and Care Excellence (NICE); 2018 Sep. Available from http://www.ncbi.nlm.nih.gov/books/NBK536075/ PMID 30645061
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Background] McMurray JJV, Packer M. How Should We Sequence the Treatments for Heart Failure and a Reduced Ejection Fraction?: A Redefinition of Evidence-Based Medicine. Circulation. 2021 Mar 2;143(9):875-877. doi: 10.1161/CIRCULATIONAHA.120.052926. Epub 2020 Dec 30. No abstract available. PMID 33378214